CLINICAL TRIAL: NCT04259008
Title: Safety of Manganese Restriction in Neonatal Parenteral Nutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Sauberan, PharmD, Clinical Research Pharmacist, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2001902
Record Dates: First submitted 2020-02-05; First posted 2020-02-06 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Infant, Newborn, Disease
Keywords: manganese, parenteral nutrition, neonate, preterm, safety
MeSH Terms: conditions — Disease; Hyperphagia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants randomized to standard trace element dose in parenteral nutrition vs. omission of manganese.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard neonatal trace elements (Active Comparator): Parenteral nutrition containing 5 mCg/kg/day manganese from "Multitrace-4 Neonatal."
  Interventions: Other: 5 mCg/kg/day manganese from "Multitrace-4 Neonatal."
- Manganese-free neonatal trace elements (Experimental): Parenteral nutrition containing the same trace element doses as "Multitrace-4 Neonatal" minus manganese.
  Interventions: Other: Manganese omission

INTERVENTIONS:
Other: Manganese omission — Participants randomized to the experimental intervention arm will not receive added manganese in their parenteral nutrition.
  Arms: Manganese-free neonatal trace elements
Other: 5 mCg/kg/day manganese from "Multitrace-4 Neonatal." — 5 mCg/kg/day manganese from "Multitrace-4 Neonatal."
  Arms: Standard neonatal trace elements

SUMMARY:
Participants will be <= 32 weeks gestational age (GA) neonates randomized to parenteral nutrition (PN) prepared with standard dose trace elements or to PN prepared with standard trace elements minus manganese.

DETAILED DESCRIPTION:
Very preterm neonates <= 32+6 weeks GA receiving PN will be randomized to receive their PN prepared with standard trace elements containing 5 mcg/kg/day of manganese, or to PN prepared with no added manganese. Randomization assignment will be double masked. All participants will have whole blood manganese measurements at baseline, at 2 weeks of postnatal age, and at 8 weeks postnatal age. Because manganese is present as a contaminant in many of the ingredients used to prepare neonatal PN, this study hypothesizes that neonates randomized to no added manganese in their PN will maintain whole blood manganese concentrations above the lower limit of normal.

ELIGIBILITY:
Inclusion Criteria:

* Inborn admissions to the SHARP Mary Birch Hospital for Women and Newborns neonatal intensive care unit.
* Less than or equal to 32+6 weeks gestational age.
* Initiated on parenteral nutrition as decided by their attending neonatologist.

Exclusion Criteria:

* Continuous exposure to routine care PN containing standard trace element for ≥ 4 hours.
* Congenital liver disease.
* Moribund status or imminent death.
* Any condition that in the judgment of the investigator or attending physician provider precludes participation because it could affect subject safety.
* Lack or refusal of informed consent

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Whole Blood Manganese | Baseline
  concentration of manganese in blood
Whole Blood Manganese | 2 weeks of age
  concentration of manganese in blood
Whole Blood Manganese | 8 weeks of age
  concentration of manganese in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jason B Sauberan, PharmD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Immediately after publication
Access Criteria: Anyone